CLINICAL TRIAL: NCT01425762
Title: Influence of Patient Choice of Intrathecal Morphine on Post-cesarean Delivery Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, Principal Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-08172011-8271; IRB 21802 (Other: Stanford University IRB)
Record Dates: First submitted 2011-08-25; First posted 2011-08-30 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Choice Group (Experimental)
  Interventions: Other: Drug Dose
- No Choice Group (Active Comparator)
  Interventions: Other: Drug Dose

INTERVENTIONS:
Other: Drug Dose — 100 versus 200 mcg IT morphine

SUMMARY:
This is a randomized controlled study that will place patients into a "choice" and a "no choice" group. The choice group will be able to choose between receiving 100 mcg or 200 mcg intrathecal morphine. The no choice group will be randomized to receive either 100 mcg or 200 mcg of intrathecal morphine. Following casarean delivery, pain scores will be measured at 3, 6, 12, 24, and 36 hours.

DETAILED DESCRIPTION:
This randomised controlled study will include pre-operative screening with a 2 simple questionnaires and the patient will be randomised into a "choice" and "no choice" groups.

The group with the choice will be offered 2 different doses of intrathecal morphine (100, 200 mcg) which they can decide on after being given a standard script explaining advantages and disadvantages of each dose. Following cesarean section patients will be followed up at 3, 6, 12, 24, 36, 48 hours following spinal injection to assess severity of pain, time to first analgesia, total analgesia requirements, treatment of nausea, vomiting and pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-50 with singleton, term gestation fetuses and scheduled for their 1st, 2nd, or 3rd elective CS (not in labor) will be included.

Exclusion Criteria:

* Patient refusal.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
pain scores (0-10) and analgesic use (morphine mg-equivalents) between the groups that have analgesic choice vs. no choice and among the actual doses received. | up to 6 months

SECONDARY OUTCOMES:
preoperative questionnaire predictor scores versus postoperative pain and analgesic consumption post cesarean delivery. | Baseline and day 1

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Carvalho B, Mirza F, Flood P. Patient choice compared with no choice of intrathecal morphine dose for caesarean analgesia: a randomized clinical trial. Br J Anaesth. 2017 May 1;118(5):762-771. doi: 10.1093/bja/aex039. PMID 28486595